CLINICAL TRIAL: NCT03019081
Title: Augmented Interoceptive Exposure Training for the Fear of Food in Anorexia Nervosa
Brief Title: Augmented Interoceptive Exposure Training in Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-013
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Isoproterenol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anorexia nervosa-study drug (Experimental): Drug: Isoproterenol Intravenous infusions of isoproterenol, delivered in a randomized double blinded order, in each participant. The isoproterenol dose will range from 0.1 micrograms to 4.0 micrograms and exposure during each visit will not exceed 25.0 micrograms. Participants will rate the experience of heartbeat and breathing sensations as well as anxiety induced by the infusion.
  Other Names: Isuprel
  Interventions: Drug: Isoproterenol
- Anorexia nervosa-placebo (Placebo Comparator): Drug: Normal Saline Intravenous infusions of normal saline, delivered in a randomized double blinded order, in each participant. Participants will rate the experience of heartbeat and breathing sensations as well as anxiety induced by the infusion.
  Other Names:
  Saline
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Isoproterenol — The goal of this experiment is to use isoproterenol in the context of inhibitory fear learning to reduce eating-related anxiety in AN, and to explore whether these changes are related to interoceptive awareness and autonomic reactivity.
  Other Names: Isuprel
  Arms: Anorexia nervosa-study drug
Other: placebo — placebo
  Other Names: Normal Saline
  Arms: Anorexia nervosa-placebo

SUMMARY:
The researchers propose to utilize a pharmacological approach involving infusions of the sympathomimetic agent isoproterenol to repeatedly trigger cardiorespiratory sensations and anxiety during meal anticipation, to facilitate the development of tolerance or a reduction of the anxiety/fear response in individuals with anorexia nervosa. The investigators aim to conduct a proof of principle study to assess for evidence of initial efficacy of this new treatment approach. As a comparator condition, the researchers propose using repeated administration of saline infusions.

DETAILED DESCRIPTION:
Individuals with anorexia nervosa (AN) are afraid to eat. Moreover, anxiety is a prominent symptom in AN, with anxiety disorders frequently preceding and/or co-occurring with the illness, and with an increased prevalence of anxiety disorders in first-degree family members. Pre-meal anxiety poses a frequent challenge in treatment settings which require adherence to strict meal plans, particularly since it is associated with lower caloric intake. While problematic under current treatment settings, this illness characteristic also provides a potentially important therapeutic target. Unfortunately, straightforward pre-meal treatment with typically effective anxiolytic medicines such as alprazolam are ineffective in individuals with AN, nor do they increase caloric intake. By contrast, cognitive behavioral therapies for anorexia nervosa utilizing exposure therapy, the most effective psychological intervention for anxiety and anxiety disorders, can promote food intake and increase weight in AN. However, such treatments are slow and have less than ideal response rates, suggesting that they could benefit from further optimization. Exposure therapy involves helping patients to voluntarily engage in repeated and sometimes prolonged confrontation with the stimulus that disproportionately provokes the individual's fear. The aim of this practice is to facilitate the development of tolerance or a reduction of the anxiety/fear response that has become conditionally associated with the relevant stimulus, thereby demonstrating to patients that they can learn to manage effectively in the face of anxiety. In the case of anorexia nervosa, the repeated presentation of food and food cues (mental imagery, pictures, smells) elicits distress and facilitates the subsequent development of tolerance of these symptoms. Unfortunately, the effect size of this intervention in AN is relatively small. Here, the researchers investigate whether the use of an acute pharmacological intervention in the context of aversive learning to enhance exposure training can reduce anxiety associated with eating in individuals with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a body mass index between 17 to 35 kg/m²
2. Must be able to provide written informed consent and must have sufficient proficiency in the English language to understand and complete interviews, questionnaires, and all other study procedures.
3. Must be capable of performing all tasks during each session of the experiment.

Inclusion criteria (AN participants, n = 50):

Participants (ages 18 to 40) must meet Diagnostic and Statistical Manual (DSM 5) criteria for Anorexia Nervosa, either current or lifetime, or have an Eating Disorder Screen (SCOFF) score ≥ 2 and a current BMI of 17 or greater. Selected medications are allowed, including selective serotonin reuptake inhibitors and benzodiazepines. Mood stabilizers and antipsychotic medications are excluded.

Exclusion Criteria:

1. No telephone or limited access to a telephone
2. Has any of the following DSM 5 disorders:

   1. Schizophrenia Spectrum and Other Psychotic Disorders
   2. Bipolar and Related Disorders
   3. Antisocial Personality Disorder
3. Active suicidal ideation with intent or plan
4. Obesity with a body mass index > 35 preventing scanner entry.
5. Illicit stimulant drugs consumed within the past week including methamphetamine or cocaine, assessed via urine drug screen
6. Active drug or alcohol dependence, or active binge drinking within the last month
7. Pregnancy as detected by a urine test
8. Prescription of a medication outside of the accepted range, as determined by best clinical practices and current research.
9. Change in the dose or prescription of a medication within the 3 weeks before enrolling in the study that could affect subjective responses, e.g., anxiolytics or antidepressants.
10. Presence of unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disease; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.
11. Non-correctable vision or hearing problems.
12. Systolic blood pressure > 160 mmHg
13. Diastolic blood pressure > 100 mmHg

Additional AN-specific exclusion criteria (AN participants):

1. Any AN individual reporting a history of cardiac or respiratory disease
2. AN with 12-lead EKG abnormalities other than bradycardia or occasional premature ventricular complexes (PVCs); those with severe bradycardia, e.g. heart rate less than 40 bpm will be excluded.
3. AN reporting a seizure within the past year
4. Active antipsychotic, mood stabilizer, lithium, stimulant, or wellbutrin medication prescription.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01; Primary Completion 2021-08 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Immediately after drug/placebo infusion
  Visual analogue self report rating scale
Sensation intensity | Immediately after drug/placebo infusion
  Heartbeat and breathing sensation intensity via self report rating scale

SECONDARY OUTCOMES:
Anxiety sensitivity index | Immediately after drug/placebo infusion
  Self report rating scale
Positive and Negative Affect | Immediately after drug/placebo infusion
  Self report rating scale
Inventory of Depression and Anxiety | Immediately after drug/placebo infusion
  Self report rating scale
Multidimensional Assessment of Interoceptive Awareness | Immediately after drug/placebo infusion
  Self report rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Sahib S Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No